CLINICAL TRIAL: NCT00046917
Title: An Open-Labeled, Non-Randomized Phase I Study of Alvocidib (Flavopiridol) Administered With Irinotecan (CPT-11) and Cisplatin in Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00023; NCI-2009-00023 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-5700; CDR0000257034; MSKCC-02043; 02-043A (Other: Memorial Sloan-Kettering Cancer Center); 5700 (Other: CTEP); P30CA008748 (NIH); R01CA067819 (NIH); U01CA069856 (NIH); NCT01645462 (obsolete NCT alias)
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2011-10

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — alvocidib; Irinotecan; Cisplatin

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients are stratified according to the number of prior treatment regimens (0 or 1 vs more than 1). Patients receive irinotecan hydrochloride IV over 30 minutes followed immediately by cisplatin IV over 30 minutes followed 7 hours later by alvocidib IV over 1-4.5 hours weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: alvocidib; Drug: irinotecan hydrochloride; Drug: cisplatin

INTERVENTIONS:
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP

SUMMARY:
Phase I trial to study the effectiveness of combining alvocidib, irinotecan hydrochloride, and cisplatin in treating patients who have advanced solid tumors. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose of flavopiridol (alvocidib), irinotecan (irinotecan hydrochloride), and cisplatin in patients with advanced solid tumors.

II. Determine the clinical pharmacokinetics of this regimen in these patients. III. Determine, preliminarily, the therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study.

Patients are stratified according to the number of prior treatment regimens (0 or 1 vs more than 1). Patients receive irinotecan hydrochloride intravenously (IV) over 30 minutes followed immediately by cisplatin IV over 30 minutes followed 7 hours later by alvocidib IV over 1-4.5 hours weekly for 2 weeks. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of cisplatin, alvocidib, and irinotecan hydrochloride until the maximum tolerated dose (MTD) of each is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 12 additional patients are treated at the recommended phase II dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic solid tumor that is refractory to standard therapy or for which no standard therapy exists
* Evaluable disease
* No previously untreated CNS metastasis
* No primary CNS tumors
* Performance status - Karnofsky 60-100%
* Performance status - ECOG 0-2
* Not specified
* WBC at least 3,000/mm^3
* Neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 2.0 mg/dL
* AST and ALT no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance at least 60 mL/min
* No cardiac arrhythmia
* No congestive heart failure
* No myocardial infarction within the past 6 months
* HIV negative
* No neuropathy grade 2 or greater
* No serious or uncontrolled infection
* No other medical condition or reason that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 2 months after study participation
* At least 4 weeks since prior immunotherapy
* At least 1 week since prior irinotecan and cisplatin alone
* At least 4 weeks since other prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* Not specified
* At least 4 weeks since prior radiotherapy
* Not specified
* Recovered from all prior therapy
* No concurrent vitamins, antioxidants, or herbal supplements except a daily multivitamin
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2002-07; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
MTD alvocidib when administered in conjunction with irinotecan hydrochloride and cisplatin | Course 1
  Defined as the dose one level below the dose at which two or more of the patients in the initial cohort experience dose limiting toxicity (DLT) during the first treatment course. DLT is defined as the occurrence of Grade 4 hematologic toxicity, Grade 3 or 4 non-hematologic toxicity including diarrhea despite antidiarrheal prophylaxis, or any delay in treatment resulting in less than 2 treatments in 3 weeks.

SECONDARY OUTCOMES:
Clinical pharmacokinetics of the regimen | Week 1 of courses 1 and 2
Therapeutic activity of alvocidib in combination with irinotecan hydrochloride in patients with advanced solid tumors | After 2 courses of treatment
  Evaluated using Response Evaluation Criteria In Solid Tumors (RECIST).
Safety and tolerability | Weekly
  Evaluated using the National Cancer Institute (NCI) Common Toxicity Criteria. Tabulated individually, and summarized by body system, according to dosage of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Shah, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States